CLINICAL TRIAL: NCT04433416
Title: Effect of Preoperative Hypertension and Controlled Hypotension on Postoperative Delirium in the Elderly
Brief Title: Hypertension and Controlled Hypotension in the Elderly
Status: Completed | Type: Observational
Sponsor: Zhang Lei (Other)
Responsible Party: Sponsor-Investigator, Zhang Lei, Deputy Chief Physician and Associate Researcher, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Organization: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Other Study IDs: SH9H-2020-T21-3
Record Dates: First submitted 2020-06-13; First posted 2020-06-16 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium | interventions — Dietary Approaches To Stop Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hypertension: After admission, two or more of the three blood pressure measurements under the same period of calm state that met hypertension, and the patient reported that he had a history of hypertension and that the blood pressure reached the standard of hypertension in the previous non-medication state was included in the hypertension group
  Interventions: Diagnostic Test: hypertension
- non-hypertension: Patients who denied the history of hypertension and were not taking antihypertensive drugs after admission and had normal blood pressure measurements were included in the non-hypertensive group

INTERVENTIONS:
Diagnostic Test: hypertension — If the patient has two or more blood pressure values ≥140/90mmHg in a calm state, he is included in this group
  Groups: hypertension

SUMMARY:
Comparision of Exposed Factors of Preoperative Hypertension and Intraoperative Controlled Hypotension on Postoperative Delirium in the Elderly under Radical Resection of Head, Neck and Maxillofacial Tumor

DETAILED DESCRIPTION:
Postoperative delirium has a higher incidence in elderly patients after general anesthesia，and It is closely related to the type of surgery, the length of surgery, and the patient's physique.Because head and neck maxillofacial radical surgery requires free flap transplantation and longer duration,and hemorrhage is more when the primary focus is removed，Intraoperative blood pressure reduction is needed to reduce bleeding，therefore, hypoperfusion of craniocerebral blood flow will occur.Low cerebral perfusion is closely related to the occurrence of postoperative delirium.Patients undergoing this type of surgery have more preoperative complications，hypertension is particularly common.Therefore, this study mainly studied the correlation between the preoperative blood pressure level and the controlled hypotension level in patients with radical head and neck and maxillofacial tumors and the incidence of postoperative delirium.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent radical anesthesia for oral and maxillofacial malignant tumors in our hospital
2. ASA grade is Ⅰ-Ⅱ
3. Patient is older than 60 years

Exclusion Criteria:

1. The patient has mental and mental disorders (eg schizophrenia, Alzheimer's disease)
2. There was severe anemia before operation (Hb<80g/L)
3. Patients had cerebral vascular complications such as cerebral infarction and lacunar infarction before operation
4. Patients who do not cooperate with this trial
5. Long-term use of sedative drugs or analgesics

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subject was a patient undergoing radical surgery for general anesthesia for mandibular and facial malignant tumors. The patients who had just been admitted to the hospital were preoperatively visited 2-3 days before the operation. According to whether the patient had a history of hypertension and the blood pressure value in the calm state after three admissions, Patients were divided into hypertensive group and non-hypertensive group.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2020-06-14 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2020-12-07 (Actual)

PRIMARY OUTCOMES:
Degree of delirium | up to three days after surgery
  From the first to the third day after surgery, the patient will be evaluated for delirium using the CAM scale.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, Doctor, Study Director — Study director
Locations (1):
- Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No